CLINICAL TRIAL: NCT06948656
Title: Study of the Impact of HYPOglycaemia on Sarcopenia in CIRrhosis
Acronym: HYPOCIR
Status: Recruiting | Type: Observational
Sponsor: Centre Hospitalier Universitaire Dijon (Other)
Responsible Party: Sponsor
Other Study IDs: MOUILLOT AFEF-AOI 2023
Record Dates: First submitted 2025-04-18; First posted 2025-04-29 (Actual); Last update posted 2025-09-16 (Actual); Status verified 2025-09

CONDITIONS: Cirrhosis
MeSH Terms: conditions — Fibrosis | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- patient: Patients with cirrhosis according to the 2021 EASL criteria
  Interventions: Other: fitting a blood glucose sensor; Other: food collection; Other: tests and questionnaires

INTERVENTIONS:
Other: fitting a blood glucose sensor — automatic, continuous collection by the blood glucose sensor for 14 days
Other: food collection — 14-day dietary record in a notebook for the patient
Other: tests and questionnaires — measurement of muscle strength using a hand-held dynamometer, animal enumeration test, self-questionnaire on the frequency of consumption of the main food groups

SUMMARY:
Fasting blood glucose is maintained by hepatic production of glucose from glycogenolysis or gluconeogenesis. In cirrhosis, glycogen storage capacity is reduced, with a consequent increase in gluconeogenesis to maintain blood glucose levels. Hypoglycaemia is particularly common during periods of prolonged nocturnal fasting. Cirrhosis can therefore be considered an 'accelerated fasting' disease. In a recent study, Honda et al. described 22% nocturnal hypoglycaemia in 105 patients analysed continuously. A previous study showed that the percentage of hypoglycaemia over the total duration of continuous blood glucose recording averaged 4%.

This gluconeogenesis could lead to a significant increase in muscle and fat catabolism, which would aggravate sarcopenia and lead to undernutrition. Undernutrition and sarcopenia are serious and severe in cirrhotic patients. Sarcopenia, present in around 45% to 67% of cirrhotic patients, is thought to lead to a significant increase in the morbidity and mortality of cirrhotic patients. Glycaemic disorders appear to play a major role in this sarcopenia. Shortening the duration of fasting, and therefore of proteolysis and lipolysis, by taking a snack in the evening, could improve nitrogen balance and glucose tolerance.

However, no study has clearly established the relationship between variations in continuous monitoring of interstitial glucose, particularly periods of nocturnal hypoglycaemia, and sarcopenia. New technologies in diabetology make it possible to obtain continuous monitoring of interstitial glucose. In addition, the use of muscle surface area at the level of the 3rd lumbar vertebra or the diameter of the psoas, obtained by scanner or MRI, combined with the use of a hand-held dynamometer to quantify muscle strength, make it easier to diagnose and assess the severity of sarcopenia and malnutrition.

The hypothesis of this work is based on the probable correlation between the time spent in hypoglycaemia (glycaemia < 0.7 g/l) and the presence of sarcopenia responsible for undernutrition in cirrhotic patients.

If positive, the results of this descriptive pilot study could provide fundamental data for anticipating and better managing sarcopenia and glycaemic disorders. The results will enable a multi-centre randomised controlled intervention trial to be set up to optimise nutritional management of patients and thus effectively combat undernutrition in cirrhotic patients.

ELIGIBILITY:
Inclusion criteria:

* Age ≥18 years
* Person with oral consent
* Patient with cirrhosis according to the 2021 EASL criteria (1)
* Patient receiving regular six-monthly and systematic monitoring of cirrhosis, according to the European recommendations of the EASL (2), or French recommendations of the TNCD (3) and HAS (4), including a clinical examination, a biological work-up (to calculate the CHILD-PUGH score and monitor alpha-feto-protein), AND requiring imaging to screen for HCC of hepatocellular carcinoma using cross-sectional imaging (by MRI and/or hepatic CT scan).

Exclusion Criteria:

* Patients with active cancer or treated within the last 6 months
* Patient with an acute episode of cirrhosis decompensation (ongoing antibiotic treatment for an active infection, gastrointestinal bleeding, hepatic encephalopathy, acute alcoholic hepatitis) less than one month old.
* Treatment with systemic corticosteroids, in progress or within the last 3 months
* Patient with organ transplant
* Person not affiliated to or not benefiting from a social security scheme
* Person under legal protection (curatorship, guardianship)
* Person subject to a legal protection measure
* Pregnant or breast-feeding women
* An adult who is incapable or unable to give consent
* Minors
* Patients already included in an interventional study who may interfere with the evaluation of this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Cirrhotic subjects will be recruited from the hepato-gastroenterology departments of the centres taking part in this clinical study.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2025-09-09 (Actual); Primary Completion 2027-10 (Estimated); Study Completion 2027-10 (Estimated)

PRIMARY OUTCOMES:
The number of nocturnal dysglycaemic events by the blood glucose sensor | For 14 days
  Defined by an episode of hypoglycaemia (blood glucose < 0.7 g/L), severe hypoglycaemia (blood glucose < 0.55 g/L) or hyperglycaemia (blood glucose > 1.8 g/L) lasting at least 15 consecutive minutes) of continuous recording of interstitial blood glucose (with Freestyle libre®). The nocturnal period is defined as the period between 11pm and 7am.
Duration of nocturnal dysglycaemic events by the blood glucose sensor | For 14 days
  Defined by an episode of hypoglycaemia (blood glucose < 0.7 g/L), severe hypoglycaemia (blood glucose < 0.55 g/L) or hyperglycaemia (blood glucose > 1.8 g/L) lasting at least 15 consecutive minutes) of continuous recording of interstitial blood glucose (with Freestyle libre®). The nocturnal period is defined as the period between 11pm and 7am.
The severity of nocturnal dysglycaemic events by the blood glucose sensor | For 14 days
  Defined by an episode of hypoglycaemia (blood glucose < 0.7 g/L), severe hypoglycaemia (blood glucose < 0.55 g/L) or hyperglycaemia (blood glucose > 1.8 g/L) lasting at least 15 consecutive minutes) of continuous recording of interstitial blood glucose (with Freestyle libre®). The nocturnal period is defined as the period between 11pm and 7am.

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Dijon Bourgogne, Dijon, France

IPD SHARING:
Plan to Share IPD: No